CLINICAL TRIAL: NCT00273910
Title: Evaluation of the Impact of Adjuvants Accompanying Peptide Immunization in High Risk Melanoma
Brief Title: Evaluation of the Impact of Adjuvants Accompanying Peptide Immunization in High-Risk Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, Dr. Steven Rosenberg, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 060069; 06-C-0069; NCT00304057 (obsolete NCT alias)
Record Dates: First submitted 2006-01-07; First posted 2006-01-09 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: High-Risk Melanoma
Keywords: Disease Free Survival; gp 100:209-217 (210m); Immunologic Response; Adjuvant Therapy; Cutaneous Melanoma; Melanoma
MeSH Terms: conditions — Melanoma | interventions — montanide ISA 51; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Adj-3 A2 gp209(2M) in IFA SQ (vortex) (Experimental): gp100:209-217(210M) peptide emulsified in MONTANIDE ISA-51 or Montanide ISA 51 VG injected subcutaneously on day one every three weeks (1 cycle) for a total of twelve cycles (33 weeks).
  Interventions: Drug: gp100:209-217 (210M); Drug: Montanide ISA-51
- Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (vortex) (Experimental): gp100:209-217(210M) peptide emulsified in MONTANIDE ISA-51 or Montanide ISA 51 VG injected subcutaneously on day one every three weeks (1 cycle) for a total of twelve cycles (33 weeks); following the injection patients will apply imiquimod to the skin at the site of injection daily for 5 days.
  Interventions: Drug: gp100:209-217 (210M); Drug: Montanide ISA-51; Drug: Imiquimod
- Adj-3 A2 gp209(2M) in saline ID (Experimental): gp100:209-217(210M) in 0.9% Sodium Chloride Injection injected intradermally on day one every three weeks (1 cycle) for a total of twelve cycles (33 weeks).
  Interventions: Drug: gp100:209-217 (210M)
- Adj-3 A2 gp209(2M) in saline ID + Imiquimod (Experimental): gp100:209-217(210M) peptide in 0.9% Sodium Chloride Injection injected intradermally on day one every three weeks (1 cycle) for a total of twelve cycles (33 weeks); following the injection patients will apply imiquimod to the skin at the site of the injection daily for 5 days.
  Interventions: Drug: gp100:209-217 (210M); Drug: Imiquimod
- Adj-3 A2 gp209(2M) in IFA SQ (2 Syringe) (Experimental): gp100:209-217(210M) peptide emulsified in Montanide ISA 51 VG injected subcutaneously on day one every three weeks (1 cycle) for a total of twelve cycles (33 weeks).
  Interventions: Drug: gp100:209-217 (210M); Drug: Montanide ISA-51
- Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (2 Syringe) (Experimental): gp100:209-217(210M) peptide emulsified in Montanide ISA 51 VG injected subcutaneously on day one every three weeks (1 cycle) for a total of twelve cycles (33 weeks); following the injection patients will apply imiquimod to the skin at the site of injection daily for 5 days.
  Interventions: Drug: gp100:209-217 (210M); Drug: Montanide ISA-51; Drug: Imiquimod

INTERVENTIONS:
Drug: gp100:209-217 (210M)
Drug: Montanide ISA-51
  Arms: Adj-3 A2 gp209(2M) in IFA SQ (2 Syringe); Adj-3 A2 gp209(2M) in IFA SQ (vortex); Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (2 Syringe); Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (vortex)
Drug: Imiquimod — Apply imiquimod 5% cream to the skin at the site of injection daily for 5 days
  Other Names: Aldara
  Arms: Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (2 Syringe); Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (vortex); Adj-3 A2 gp209(2M) in saline ID + Imiquimod

SUMMARY:
This study will evaluate the immunization effects of a vaccine for patients who are at risk for recurrence of their skin cancer. That is, the risk of cancer is higher if melanoma has invaded deep into the skin or lymph nodes. Currently, the only therapy that the U.S. Food and Drug Administration (FDA) has approved for preventing recurrence of melanoma is alpha-interferon. But the research data are controversial. In this study, the vaccine to be used, called gp100, contains a piece of a protein called a peptide, which melanoma cancer cells produce.

Patients 16 and older who have had confirmed melanoma surgically removed and whose tissue type is tested as being human leukocyte antigen serotype within HLA-A serotype group (HLA-A2), through a specific blood test, may be eligible for this study.

Up to 132 participants will be enrolled. There will be a physical examination and collection of blood samples for tests, and making sure that x-rays and scans are current. Patients will be randomly assigned to four groups. Group 1 will receive the peptide with an adjuvant (assistant) oil-based liquid called Montanide ISA-51, as an injection in the thigh. Group 2 will receive gp100, Montanide, and a cream called imiquimod, which the FDA has approved for treating genital warts and herpes but that may help immune cells in the skin to recognize the vaccine. Imiquimod will be applied to the skin for 5 days. Group 3 will receive gp100 mixed in salt water given as several mini-doses under the skin of the thigh. Group 4 will also receive several mini-doses of gp100 mixed in saline, as well as imiquimod cream applied to the skin for 5 days. All patients will receive the gp100 every 3 weeks for 12 weeks. Every dose is a cycle, with four cycles considered a course of therapy. If the melanoma does not return or patients do not experience side effects from this therapy, then the courses of vaccine will repeated for up to 12 cycles of therapy (3 courses over 33 weeks). Side effects of the peptide vaccination include local swelling, swelling of local lymph nodes, bruising, and pain and redness at the injection sites. There may be chills or fever. Patients will be watched closely for such side effects.

To study how the vaccine changes the action of cells in the immune system, patients' white blood cells (lymphocytes) will be obtained, involving a separate informed consent. The procedure, called leukaphersis, requires inserting a needle into the arm, to obtain blood going into a machine, which divides the blood into red cells, plasma (or the serum part), and lymphocytes. The lymphocytes are removed, and the plasma and red cells returned to the patient through a second needle in the other arm. Risks associated with the procedure include fainting, which can be prevented by patients' eating before coming to the lab, and bleeding and infection at the needle site. Patients will undergo leukapheresis will be done about four times: before receiving the vaccine, 3 weeks after the first four doses, and then after 8 cycles and 12 cycles. Patients assigned to the groups receiving imiquimod will be asked to record every time they apply that cream and describe any symptoms developed during the study. All patients will be watched closely for any sign that their melanoma has returned. Before and throughout the study, multiple blood tests will be conducted.

The vaccine, Montanide, and imiquimod may increase patients' immune system in fighting off new tumors, but that is not known now. However, the study may provide information that will be useful in treating melanoma patients in the future.

DETAILED DESCRIPTION:
Background:

A previous clinical trial has been conducted in the Surgery Branch National Cancer Institute (NCI) in which gp100 immunizations have been administered to patients with melanoma in the adjuvant setting. In this prior protocol, the peptide emulsified in Incomplete Freund's Adjuvant was administered subcutaneously using several different schedules and was well tolerated except for mild and transient erythema at the site of injection. Each of the schedules provided successful immunization although the q3w schedule was the best tolerated locally and three courses of immunization appeared to be sufficient using this regimen. An important finding from the adjuvant protocol however was the significant increase in immune precursors specifically reactive against peptide and tumor that occurred with increasing courses of immunization. These findings have encouraged us to now further explore the optimal methods for generating immune precursors using the gp100:209-217(210M) peptide by testing the impact of an additional immune adjuvant, imiquimod, reported to increase the immunizing potential of antigens as well as evaluate an alternate route of injection, intradermal administration.

Objectives:

The primary objective of this trial is to evaluate the immunologic activity of immunization with four different preparations of the gp100:209-217(210M) melanoma antigen peptide and potentially select one for further study.

Eligibility:

HLA-A 0201 patients, age greater than or equal 16 years, with primary melanomas with lesions that are ulcerated and greater than or equal 2mm, or any lesions that are greater than or equal 4.0 mm in thickness, or greater than or equal 1 positive lymph node, or local recurrence, or resected metastatic disease, within 6 months of surgical resection will be considered. Patients who have ocular or mucosal melanoma or who require systemic steroid therapy will be excluded. The following patients will also be excluded: have previously been immunized with gp100; have known hypersensitivity to any of the agents used in this study; have previously received chemotherapy for treatment of melanoma; or who are undergoing or have undergone in the past 3 weeks any systemic therapy except surgery for their cancer.

Design:

Patients will be randomized into one of the following four arms:

1. gp100:209-217(210M) peptide emulsified in MONTANIDE ISA-51 or Montanide ISA 51 VG injected subcutaneously on day one every three weeks (1 cycle) for a total of twelve cycles (33 weeks).
2. gp100:209-217(210M) peptide emulsified in MONTANIDE ISA-51 or Montanide ISA 51 VG injected subcutaneously on day one every three weeks (1 cycle) for a total of twelve cycles (33 weeks); following the injection patients will apply imiquimod to the skin at the site of injection daily for 5 days.
3. gp100:209-217(210M) in 0.9% Sodium Chloride Injection injected intradermally on day one every three weeks (1 cycle) for a total of twelve cycles (33 weeks).
4. gp100:209-217(210M) peptide in 0.9% Sodium Chloride Injection injected intradermally on day one every three weeks (1 cycle) for a total of twelve cycles (33 weeks); following the injection patients will apply imiquimod to the skin at the site of the injection daily for 5 days.

Immunizations will be administered on an outpatient basis unless side effects or the patient's clinical condition warrants hospitalization. Patients will receive full clinical evaluation three weeks after 8 cycles and 12 cycles.

Each of the arms will be conducted using a two-stage optimal design Since the primary objective is to select one regimen from among the four on the basis of the immune response, this design allows there to be greater than 80% probability of correctly selecting the superior arm if there is either a tie in the number of immune responses, or if there is at least one more immune response on one arm than the other three arms, and if the true response rates are 15%, 15%, 15% and 35%. Initially, 19 patients will be enrolled in each arm and evaluated; if 0 to 3 of 19 in an arm have an immune response to T2 cells pulsed with 0.01 M peptide after the 4th, 8th, and 12th cycles, no further patients would be randomized to receive the peptide on that arm. If at least four immunologic responses are noted after the 8th cycle, then accrual to 33 patients would take place. If all four arms need to be completed and 33 patients need to be completed in each arm, a total of 132 patients are required.

ELIGIBILITY:
* INCLUSION CRITERIA:

HLA-A 0201 patients, age greater than or equal to 16 years, primary melanomas with lesions that are ulcerated and greater than or equal to 2mm, or any lesions that are greater than or equal to 4.0 mm in thickness, or greater than or equal to1 positive lymph node, or local recurrence, or resected metastatic disease, within 6 months of surgical resection will be considered. Patients must be clinically disease free at the time of protocol entry as documented by radiologic studies within 6 weeks of patient entry.

Serum creatinine of 2.0 mg/dl or less

Total bilirubin 1.6 mg/dl or less, except for patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.

WBC 3000/mm^3 or greater,

Platelet count 90,000 mm^3 or greater,

Serum aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than three times normal,

Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Patients of both genders must be willing to practice effective birth control during this trial because the potential for teratogenic effects are unknown.

Patients may have had prior adjuvant treatment with immunotherapy, including interferon, as long as 3 weeks have elapsed since prior systemic therapy.

EXCLUSION CRITERIA:

Patients will be excluded:

Who have ocular or mucosal melanoma.

Who are undergoing or have undergone in the past 3 weeks any systemic therapy except surgery for their cancer, and must have recovered to a grade I from any adverse effects of treatment prior to entry, other than those that do not have clinical implications, e.g. vitiligo, alopecia.

Have active systemic infections, autoimmune disease or any known immunodeficiency disease.

Who require systemic steroid therapy.

Who are pregnant (because of possible side effects on the fetus) or breastfeeding because of unknown effects on the developing child).

Who are known to be positive for hepatitis BsAG or human immunodeficiency virus (HIV) antibody (because of possible immune effects of these conditions).

Who have any form of autoimmune disease (such as autoimmune colitis or Crohn's Disease) or immunodeficiency as evidenced by abnormal white blood count (WBC) count 8 and/or presence of opportunistic infections. Must have recovered immune competence after radiation therapy. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)

Who have previously been immunized with gp100.

Who have known hypersensitivity to any of the agents used in this study.

Who have previously received chemotherapy for treatment of melanoma.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2006-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kawakami Y, Eliyahu S, Delgado CH, Robbins PF, Rivoltini L, Topalian SL, Miki T, Rosenberg SA. Cloning of the gene coding for a shared human melanoma antigen recognized by autologous T cells infiltrating into tumor. Proc Natl Acad Sci U S A. 1994 Apr 26;91(9):3515-9. doi: 10.1073/pnas.91.9.3515. PMID 8170938
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2006-C-0069.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 104 subjects were enrolled in this trial.
Period: Overall Study
Arm/Group | Adj-3 A2 gp209(2M) in IFA SQ (Vortex) | Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (Vortex) | Adj-3 A2 gp209(2M) in Saline ID | Adj-3 A2 gp209(2M) in Saline ID + Imiquimod | Adj-3 A2 gp209(2M) in IFA SQ (2 Syringe) | Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (2 Syringe)
Started | 19 | 19 | 18 | 19 | 15 | 14
Completed | 19 | 19 | 18 | 19 | 15 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adj-3 A2 gp209(2M) in IFA SQ (Vortex) | Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (Vortex) | Adj-3 A2 gp209(2M) in Saline ID | Adj-3 A2 gp209(2M) in Saline ID + Imiquimod | Adj-3 A2 gp209(2M) in IFA SQ (2 Syringe) | Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (2 Syringe) | Total
Number analyzed (Participants) | 19 | 19 | 18 | 19 | 15 | 14 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 18 | 19 | 13 | 14 | 102
  >=65 years | 0 | 0 | 0 | 0 | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 46.9 (9.1) | 42.8 (10.4) | 48.8 (12.7) | 48.1 (10.2) | 51.7 (13.2) | 47.7 (8.3) | 47.6 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 9 | 6 | 3 | 4 | 37
  Male | 13 | 10 | 9 | 13 | 12 | 10 | 67
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaskan Natives | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian or Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black of non-Hispanic Origin | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hispanic | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White of non-Hispanic Origin | 18 | 19 | 18 | 19 | 15 | 14 | 103
  Other or Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 18 | 19 | 15 | 14 | 104

OUTCOME MEASURES:

1. Primary Outcome: Immunologic Response Rate
Description: Comparison of six different preparations of the gp100:209-217 (210M) melanoma antigen peptide. The arm with the greater number of immunologic responses will be the one most likely to be selected for future study on the basis of immunization alone. Evidence of immunization consist of at least 10 Elispots/100,000 cells above background. An injection site reaction is not an immune response.
Time Frame: 48 months
Population: The number of participants analyzed and results are correct. We do not have the immunologic response rate data for all patients.
Measure: Number; unit: Participants
Arm/Group | Adj-3 A2 gp209(2M) in IFA SQ (Vortex) | Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (Vortex) | Adj-3 A2 gp209(2M) in Saline ID | Adj-3 A2 gp209(2M) in Saline ID + Imiquimod | Adj-3 A2 gp209(2M) in IFA SQ (2 Syringe) | Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (2 Syringe)
Number analyzed (Participants) | 14 | 10 | 12 | 15 | 5 | 5
Participants | 2 | 0 | 0 | 3 | 1 | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 48 months
Measure: Number; unit: Participants
Arm/Group | Adj-3 A2 gp209(2M) in IFA SQ (Vortex) | Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (Vortex) | Adj-3 A2 gp209(2M) in Saline ID | Adj-3 A2 gp209(2M) in Saline ID + Imiquimod | Adj-3 A2 gp209(2M) in IFA SQ (2 Syringe) | Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (2 Syringe)
Number analyzed (Participants) | 19 | 19 | 18 | 19 | 15 | 14
Participants | 19 | 19 | 18 | 19 | 15 | 14

ADVERSE EVENTS:
Time Frame: 48 months
Arm/Group | Adj-3 A2 gp209(2M) in IFA SQ (Vortex) | Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (Vortex) | Adj-3 A2 gp209(2M) in Saline ID | Adj-3 A2 gp209(2M) in Saline ID + Imiquimod | Adj-3 A2 gp209(2M) in IFA SQ (2 Syringe) | Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (2 Syringe)
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/18 | 0/19 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 19/19 | 19/19 | 18/18 | 19/19 | 15/15 | 14/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adj-3 A2 gp209(2M) in IFA SQ (Vortex) (N=19) | Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (Vortex) (N=19) | Adj-3 A2 gp209(2M) in Saline ID (N=18) | Adj-3 A2 gp209(2M) in Saline ID + Imiquimod (N=19) | Adj-3 A2 gp209(2M) in IFA SQ (2 Syringe) (N=15) | Adj-3 A2 gp209(2M) in IFA SQ + Imiquimod (2 Syringe) (N=14)
Leukocyte count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sweating (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 19 (56) | 19 (48) | 18 (47) | 19 (55) | 15 (35) | 14 (36)
Pruritis (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No